CLINICAL TRIAL: NCT04308330
Title: A Phase I Study of Vorinostat in Combination With Vincristine, Irinotecan, and Temozolomide in Children, Adolescents, and Young Adults With Relapsed or Refractory Solid Tumors and CNS Malignancies
Brief Title: Vorinostat in Combination With Chemotherapy in Relapsed/Refractory Solid Tumors and CNS Malignancies
Acronym: NYMC195
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12011
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Ewing Sarcoma; Rhabdomyosarcoma; Wilms Tumor; Neuroblastoma; Hepatoblastoma; Germ Cell Tumor
MeSH Terms: conditions — Sarcoma, Ewing; Rhabdomyosarcoma; Wilms Tumor; Neuroblastoma; Hepatoblastoma; Neoplasms, Germ Cell and Embryonal | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vorinostat (Experimental): The first cycle of chemotherapy will not include the experimental agent vorinostat. This first cycle will be used to determine whether the patient can tolerate the chemotherapeutic backbone without developing a DLT.
  Cycle 1
  * Vincristine: 1.5 mg/m2/day (maximum dose 2 mg) IV Days 1 and 8 over 1-15 minutes.
  * Temozolomide: 125 mg/m2/day PO Days 1-5.
  * Irinotecan: 50 mg/m2/day IV Days 1-5 over 60 minutes.
  * Cefixime: 8 mg/kg/day (maximum dose 400 mg) PO. Begin 2 days prior to irinotecan therapy and continue through Day 8.
  Cycles 2-12
  * Vincristine: 1.5 mg/m2/day (maximum dose 2 mg) IV Days 1 and 8 over 1-15 minutes.
  * Temozolomide: 125 mg/m2/day PO Days 1-5.
  * Irinotecan: 50 mg/m2/day IV Days 1-5 over 60 minutes.
  * Cefixime: 8 mg/kg/day (maximum dose 400 mg) PO. Begin 2 days prior to irinotecan therapy and continue through Day 8.
  * Vorinostat: Dose per escalation schema daily Days 1-5.
  * Vorinostat will not be administered during Cycle 1.
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — This is a phase I study of the combination of four drugs: vorinostat, vincristine, irinotecan, and temozolomide. This is called a Phase I study because the goal is to find the highest dose of vorinostat that investigators can give safely when it is used together with the chemotherapy drugs vincristine, irinotecan and temozolomide. Investigators are using vorinostat because it seems to work against cancer in test tubes and animals. It may be most effective when it is given with chemotherapy. The combination of these three agents together has never been given to children. Vincristine, irinotecan, and temozolomide are approved and used for the treatment of other types of cancer in adults and children. Vorinostat is approved and used to treat cancer in adults. The combination of these four drugs together is experimental. Investigators do not know if this combination of medicines will work in people. There is a lot that investigators do not yet know about this combination of medicines.
  Other Names: Zolinza

SUMMARY:
Investigators are testing new experimental drug combinations such as the combination of vorinostat, vincristine, irinotecan, and temozolomide in the hopes of finding a drug that may be effective against tumors that have come back or that have not responded to standard therapy.

The goals of this study are:

* To find the highest safe dose of vorinostat that can be given together with vincristine, irinotecan, and temozolomide without causing severe side effects;
* To learn what kind of side effects this four drug combination can cause;
* To learn about the effects of vorinostat and the combination of vorinostat, vincristine, irinotecan, and temozolomide on specific molecules in tumor cells;
* To determine whether the combination of vorinosat, vincristine, irinotecan, and temozolomide is a beneficial treatment.

DETAILED DESCRIPTION:
This first cycle will be used to determine whether the patient can tolerate the chemotherapeutic backbone without developing a DLT. The baseline disease evaluation will be obtained following hematologic recovery from the first cycle of chemotherapy, after which combination therapy with vorinostat will be given in subsequent cycles (2-12) w/ modifications if needed. Vorinostat dose escalation in subsequent patient cohorts will occur based on DLT to determine a MTD.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients must be less than or equal to 1 year and less than or equal to 30 years of age at initiation of protocol therapy.
* Diagnosis: Patients must have a confirmed histologic diagnosis of a relapsed or refractory solid tumor or CNS malignancy.
* Performance status: Patients over 16 years of age must have a Karnofsky score greater than or equal to 50. Children under 16 years of age must have a Lansky score greater than or equal to 50.
* Prior therapy: Patients may have received prior therapy with vincristine, irinotecan, or temozolomide. They may not however have received therapy that included a treatment cassette of irinotecan and temozolomide in combination.

  * Prior myelosuppressive therapy: Patients must have not received myelosuppressive therapy in 3 weeks or nitrosourea chemotherapy within 6 weeks of initiation of protocol therapy.
  * Hematologic growth factor support: Patients may not have received G-CSF within the previous 3 days or peg-filgrastim within the past 7 days.
  * Biologic anti-neoplastic therapy: At least 21 days or 5 half-lives (whichever is of longer duration) must have elapsed since the last administration of biologic antineoplastic therapy.
  * Radiation therapy: ≥ 14 days since the last dose of local XRT; ≥ 6 months must have elapsed if prior TBI, craniospinal XRT or ≥ 50% radiation of pelvis; ≥ 6 wks must have elapsed if other substantial BM radiation.
  * Autologous or allogeneic stem cell transplant: No active graft vs. host disease or need for immunosuppressive therapy. At least 3 months must have passed since neutrophil engraftment.
* Organ function:

Bone marrow function:

* Peripheral absolute neutrophil count (ANC) greater than or equal to 1000 cells/mcL.
* Platelet count greater than or equal to100,000/mcL and no platelet transfusion within prior 7 days.
* Hemoglobin greater than or equal to 8 gm/dL
* Patients with known bone marrow metastatic disease may enroll on the study if they have a peripheral ANC greater than or equal to 750 cells/mcL. They will not be evaluable for hematologic toxicity.

  - Adequate liver function:
* Total bilirubin less than or equal to 1.5x upper limit of normal (ULN) for age.
* SGPT (ALT) less than or equal to 5x ULN
* Serum albumin greater than or equal to 2 gm/dL

  - Adequate renal function:
* Creatinine clearance or glomerular filtration rate >70 ml/min/1.73 m2 or a serum creatinine based on age and gender as follows:

Age Maximum serum creatinine concentration (mg/dL) Male Female 1-<2 years 0.6 0.6 2-<6 years 0.8 0.8 6-<10 years 1 1 10-<13 years 1.2 1.2 13-<16 years 1.5 1.4 greater than or equal to 16 years 1.7 1.4 The threshold creatinine values in this table were derived from the Schwartz formula to estimate glomerular filtration rates (Schwartz et al. J. Peds. 106; 522. 1985) using child length and stature data from the CDC.

- Informed consent: All patients less than 18 years of age must sign a written informed consent. For patients <18 years of age, a parent or guardian must sign a written informed consent, unless the patient is an emancipated minor. Childhood assent, when appropriate, should be obtained as well per institutional guidelines.

Exclusion Criteria:

* Pregnancy or breast feeding: Women who are pregnant or breast feeding will not be entered on the protocol due to the risks of fetal and teratogenic adverse events with the therapeutic agents used in the protocol therapy.
* Corticosteroid use: Patients with CNS tumors who have not been on a stable or decreasing dose of corticosteroids for the 7 days prior to the initiation of protocol therapy.
* Antineoplastic therapy: Patients receiving any other antineoplastic therapy.
* Medication allergy:

Allergy or intolerance to any of the protocol agents: vincristine, irinotecan, temozolomide, or vorinostat.

Allergy or intolerance to cephalosporins.

* Infection: Patients who have any uncontrolled infection, positive blood culture within 48 hours prior to protocol entry, or diagnosed or receiving therapy for Clostridium difficile infection.
* Patients may not have taken valproic acid or any other histone deacetylase inhibitor for at least 2 weeks prior to study enrollment.
* Children with neurofibromastosis Type 1, if being used for treatment of a low grade glioma.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-17 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine a maximally tolerated (or optimal) dose of vorinostat | 1 year
  A minimum of 3 evaluable patients will be entered at each dose level. If no significant dose limiting toxicity is discovered, a maximum of 3 dose levels will be evaluated. The minimum patient enrollment will be 3 patients. Many of the patients enrolled on this trial are expected to be heavily pretreated. All patients will be given a VIT only "window" to evaluate adequate bone marrow reserve to tolerate protocol therapy. We expect that at most 20% of patients will not be able to tolerate VIT or VIT with dose reduced temozolomide. A maximum of 24 patients enrolled on study is anticipated. Once the MTD has been defined, up to 6 additional patients may be enrolled to acquire additional safety data regarding this combination of agents.

SECONDARY OUTCOMES:
Overall response rate (ORR) after therapy | 1 year
  To determine the overall response rate (ORR) of vorinostat in combination with VIT in children, adolescents, and young adults with relapsed or refractory solid tumors.
  The overall (CR+PR) and best response rates with the 95% confidence intervals will be estimated based on the exact binomial distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Rosenblum, MD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: No